CLINICAL TRIAL: NCT07272382
Title: Effect of Omega-3 Fatty Acids on PD-1 Inhibitor Therapy in Advanced Esophageal Cancer (ESO-Shanghai28): A Phase II Randomized Controlled Trial
Brief Title: Omega-3 Fatty Acids With PD-1 Inhibitors in Advanced Esophageal Cancer
Acronym: ESO-Shanghai28
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, MD, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESO-Shanghai28
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 + Omega-3 (EPA/DHA) (Experimental)
  Interventions: Dietary Supplement: PD-1 + Omega-3 Fatty Acids (EPA/DHA)
- PD-1 + Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: PD-1 + Placebo (Oral Drops)

INTERVENTIONS:
Dietary Supplement: PD-1 + Omega-3 Fatty Acids (EPA/DHA) — Intervention: Omega-3 (EPA 2.5 g + DHA 1.25 g/day) oral drops × 6 months; with PD-1; blinded; adherence via check-ins/bottle counts/plasma EPA/DHA.
  Arms: PD-1 + Omega-3 (EPA/DHA)
Dietary Supplement: PD-1 + Placebo (Oral Drops) — Comparator: Matching placebo oral drops × 6 months; with PD-1; blinded; adherence via check-ins/bottle counts.
  Arms: PD-1 + Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase II clinical trial designed to evaluate whether adding omega-3 fatty acids improves outcomes in adult patients with recurrent or metastatic esophageal cancer receiving PD-1 inhibitor therapy.

The main questions are:

Compared with placebo, does omega-3 (EPA+DHA) increase the longitudinal change in skeletal muscle index (ΔSMI) over 6 months? Does it improve clinical outcomes and favorably modulate immune and metabolic biomarkers as well as patient-reported outcomes ?

Participants will be randomized 1:1 to:

Intervention: Standard PD-1 therapy plus oral omega-3 (EPA 2.5 g + DHA 1.25 g per day) for 6 months.

Control: Standard PD-1 therapy plus matching placebo for 6 months. Participants will attend study visits at baseline, 3 months, and 6 months (then every 3 months up to 2 years), undergo body composition and functional assessments, blood sampling, and questionnaires, and have treatment adherence assessed per protocol. Pre-specified exploratory biomarker analyses will be conducted to support mechanism research.

ELIGIBILITY:
Inclusion Criteria： Age ≥18 years; ECOG 0-2. Histologically confirmed recurrent/metastatic esophageal cancer (AJCC 8th; de novo stage IV or relapse after prior therapy).

PD-1 inhibitor naïve, or prior PD-1 stopped >3 months with subsequent progression (not primary PD-1 resistance).

Adequate organ function per protocol (hematologic, hepatic, renal). Women of childbearing potential: negative pregnancy test and agree to effective contraception.

Signed informed consent.

Exclusion Criteria： PD-1 inhibitor resistance or refractory disease to prior PD-1. Esophageal fistula present or strongly suspected. Active autoimmune disease or immunodeficiency requiring systemic therapy (protocol-defined exceptions allowed, e.g., treated hypothyroidism; controlled type 1 diabetes).

Systemic corticosteroids or other immunosuppressants requiring ongoing use (physiologic or topical steroids allowed).

Interstitial lung disease/pneumonitis history or active pneumonitis on screening CT.

Uncontrolled cardiovascular disease (e.g., NYHA ≥ II heart failure, unstable angina, recent MI, significant uncontrolled arrhythmias).

Serious active infection, including active TB; uncontrolled viral hepatitis (active HBV/HCV per protocol).

Pregnant or breastfeeding. Recent major surgery (per protocol window) or high bleeding risk/therapeutic anticoagulation not suitable for omega-3 use.

Other conditions that, in investigator's judgment, preclude protocol compliance or safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2027-06-05 (Estimated); Study Completion 2027-06-05 (Estimated)

PRIMARY OUTCOMES:
Change in Skeletal Muscle Index (ΔSMI) From Baseline to 6 Months | From randomization to Month 6 (±4 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary publication will be shared with qualified researchers for legitimate scientific purposes. Data will be de-identified per HIPAA and local regulations.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 12 months after primary results publication and for 5 years thereafter.
Access Criteria: Researchers must submit a methodologically sound proposal, IRB/ethics approval (or exemption), and a signed data use agreement. Proposals will be reviewed by the sponsor/investigator committee.
URL: https://www.shca.org.cn/